CLINICAL TRIAL: NCT00562783
Title: A Phase II, Double-blinded, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Vitalliver in Patients With Decompensated Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Vigconic (International) Ltd. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UW04-223 T/545; HARECCTR0500001
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis B; Hepatitis C; Liver Cirrhosis
Keywords: HBV; HCV; Liver cirrhosis
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Liver Cirrhosis

INTERVENTIONS:
Drug: Vitaliver
Drug: Placebo

SUMMARY:
Cirrhosis is a diffuse lesion characterized by architectural distortion of the liver because of collagen deposition and development of nodules of regenerating hepatocytes. It is an irreversible change that results from diseases characterized by chronic liver injury (Fujimoto, 2000). Cirrhosis alters the pattern of blood flow through the liver and results in impaired perfusion of hepatic lobules with intrahepatic and extrahepatic shunting of blood. This deprives hepatocytes of uniform perfusion by arterial and portal venous blood resulting in both portal hypertension and other consequences of cirrhosis including impaired protein synthesis and altered drug metabolism. The histologic diagnosis of cirrhosis requires the presence of regenerative nodules or pseudolobules completely encircled by fibrosis such as congenital hepatic fibrosis can result in portal hypertension in the absence of cirrhosis (Anthony et al., 1977).

The events leading to the development of cirrhosis are generally those of chronic injury with hepatocyte destruction. Acute severe liver injury as in fulminant viral hepatitis does not result in cirrhosis and the liver generally returns to normal after recovery. Cirrhosis can be classified by macroscopic appearance, by cause, and by histologic appearance and location of liver damage. Micronodular cirrhosis is composed of uniform nodules less than 3 mm in diameter, whereas macronodular cirrhosis has varying size nodules greater than 3 mm diameter. Mixed nodular cirrhosis has nodules of both sizes. Some liver diseases such as alcoholic liver disease may present as micronodular cirrhosis and develop larger nodules with subsequent regeneration of hepatocytes. For this reason, many prefer etiologic classification (e.g., alcoholic cirrhosis). The designation of cirrhosis as post necrotic, biliary and portal are still commonly used and imply predominant histologic location of fibrosis.

Cirrhosis is an irreversible disease, and attempts should be made to stabilize the patient and to control the cause. Factors that indicate a poor outcome include an elevated prothrombin time that does not correct itself with parenteral vitamin K, upper gastrointestinal bleeding caused by varices, ascites refractory to therapy, increased age of the patient, sever malnutrition, spontaneous bacterial peritonitis, a pronounced increase of serum bilirubin in the absence of haemolysis, and heptocellular carcinoma (Yeh et al., 2003). In general, all causes of upper GI bleeding are associated with an increased mortality in patients with cirrhosis. For those with alcoholic cirrhosis who lack portal hypertension, survival is similar to an age-matched cohort if alcohol intake is stopped (Nakamura et al., 1991). If ethanol consumption continues, mortality is higher. Cirrhosis can be present without clinically significant complications and be identified only at autopsy or during evaluation of abnormal liver tests (Mendez et al., 2003). However, for many patients the disease is slowly progressive resulting in one or more complications. The clinical manifestations of cirrhosis are a result of altered hepatic blood flow through the liver with intrahepatic shunting causing impaired perfusion of hepatocytes or portal hypertension with shunting of blood around the liver though portosystemic communications. The major complications of portal hypertension include oesophageal or gastric varices, ascites, portosystemic encephalopathy, and hepatorenal-syndrome (Menon & Kamath, 2000). With impairment of hepatocyte perfusion or reduction of hepatocyte number, altered synthetic function can result in hypoalbuminemia, hypoprothrombinemia, and changes in drug metabolism.

Vitalliver is a Chinese medicine which is administered in the form of a suppository, which is uncommon for most Chinese medicines. Medications released from the suppositories are absorbed directly from the circulation around the rectum and then reach the liver via the portal vein.

Basic pharmacological studies have shown that Vitalliver has good immunomodulating functions, increases the activities of T-cells, B-cells and NK cells, therefore this formulation may have special values in treating liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* HBV or HCV related liver cirrhosis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-01; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome for evaluating the clinical efficacy of Vitalliver is the Model for End Stage Liver Disease (MELD) score | week 16

SECONDARY OUTCOMES:
Child-Pugh's grading | Week 16
Quality of life variable | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, Dr, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China